CLINICAL TRIAL: NCT02615301
Title: Intake of Dietary Vitamin D and K From Tailor-made Atlantic Salmon and Bone Health - A Randomized Intervention Study
Brief Title: Dietary Intake of Salmon and Bone Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Nutrition and Seafood Research, Norway (Other Government)
Collaborators: Haukeland University Hospital (Other)
Responsible Party: Principal Investigator, Jannike Øyen, Jannike Øyen, PhD, National Institute of Nutrition and Seafood Research, Norway
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 252.07
Record Dates: First submitted 2015-11-18; First posted 2015-11-26 (Estimated); Last update posted 2015-11-26 (Estimated); Status verified 2015-11

CONDITIONS: Osteoporosis
MeSH Terms: conditions — Osteoporosis | interventions — Vitamin D; Calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Salmon (HD+HK) (Experimental): Tailor-made salmon with high levels of vitamin D3 and K1
  Interventions: Dietary Supplement: Tailor-made salmon with high levels of vitamin D3 and K1
- Salmon (LD+HK) (Experimental): Tailor-made salmon with low levels of vitamin D3 and high K1
  Interventions: Dietary Supplement: Tailor-made salmon with low levels of vitamin D3 and high K1
- Salmon (HD+LK) (Experimental): Tailor-made salmon with high levels of vitamin D3 and low K1
  Interventions: Dietary Supplement: Tailor-made salmon with high levels of vitamin D3 and low K1
- Supplement (vitamin D + Calcium) (Experimental): Supplement with vitamin D and Calcium
  Interventions: Dietary Supplement: Supplement with vitamin D and Calcium

INTERVENTIONS:
Dietary Supplement: Tailor-made salmon with high levels of vitamin D3 and K1 — The aims were to investigate how intake of tailor-made salmon with high levels of vitamin D3 and K1 affected bone biomarkers, nutritional status (vitamin D, omega-3), as well as body composition and bone mineral density.
  Arms: Salmon (HD+HK)
Dietary Supplement: Tailor-made salmon with low levels of vitamin D3 and high K1 — The aims were to investigate how intake of tailor-made salmon with low levels of vitamin D3 and high K1 affected bone biomarkers, nutritional status (vitamin D, omega-3), as well as body composition and bone mineral density.
  Arms: Salmon (LD+HK)
Dietary Supplement: Tailor-made salmon with high levels of vitamin D3 and low K1 — The aims were to investigate how intake of tailor-made salmon with high levels of vitamin D3 and low K1 affected bone biomarkers, nutritional status (vitamin D, omega-3), as well as body composition and bone mineral density.
  Arms: Salmon (HD+LK)
Dietary Supplement: Supplement with vitamin D and Calcium — The aims were to investigate how supplement with vitamin D and Calcium affected bone biomarkers, nutritional status (vitamin D, omega-3), as well as body composition and bone mineral density.
  Arms: Supplement (vitamin D + Calcium)

SUMMARY:
The aims of this study were to investigate how intake of tailor-made salmon affected bone biomarkers, nutritional status, as well as body composition and bone mineral density. The 122 healthy postmenopausal women included in this 12 weeks intervention study were randomized into four groups: three salmon groups (with three different vitamin D3/vitamin K1 combinations) and one tablet group (vitamin D and Calcium).

DETAILED DESCRIPTION:
Suboptimal vitamin D status is common among humans, and might have a negative impact on bone health. Fatty fish, including Atlantic salmon, is an important dietary vitamin D source. However, due to a considerable change in fish feed composition, the contribution of vitamin D from salmon fillet has been reduced. The aims were to investigate how intake of tailor-made salmon affected bone biomarkers, nutritional status (vitamin D, omega-3), as well as body composition and bone mineral density (BMD). The 122 healthy postmenopausal women (median 55 years) included in this 12 weeks intervention study were randomized into four groups: three salmon groups (150 grams/two times/week) and one tablet group (800IU vitamin D and 1000 mg Calcium/day). The salmon groups also received calcium supplements (1000 mg/d). The salmon had three different vitamin D3/vitamin K1 combinations: high D3 + high K1, low D3 + high K1, or high D3 + low K1.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women
* Caucasian ethnicity
* Age range 50-65 years
* Having postmenopausal age of at least one year

Exclusion Criteria:

* Osteoporotic fractures
* Medical treatment for osteoporosis
* Warfarin treatment
* Creatinine above or below normal range
* Hypervitaminosis D
* Malabsorption syndrome
* Inflammatory bowel disease
* Inflammatory rheumatic diseases
* Women who had planned to go away on holiday during the intervention could not participate

Ages: 50 Years to 64 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 122 (Actual)
Dates: Start 2009-01; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Bone-specific alkaline phosphatase | 3 months
  Serum (µg/l)
Osteocalcin | 3 months
  Serum (ng/ml)
Undercarboxylated osteocalcin (GLU) | 3 months
  Serum (ng/ml)
Carboxylated osteocalcine (GLA) | 3 months
  Serum (ng/ml)
GLU/GLA-ratio | 3 months
  Ratio of undercarboxylated osteocalcin and carboxylated osteocalcine
N-telopeptides/creatinine | 3 months
  Urinary (mmol/l)
Deoxypyridinoline/creatinine | 3 months
  Urinary (mmol/l)

SECONDARY OUTCOMES:
25-hyroxyvitamin D | 3 months
  Serum 25(OH)D (nmol/L)
Eicosapentaenoic acids | 3 months
  Fatty acids composition of total red blood cells
Docosahexaenoic acids | 3 months
  Fatty acids composition of total red blood cells
Omega-3 index | 3 months
  The content of Eicosapentaenoic acids and Docosahexaenoic acids in red blood cell membranes expressed as percent of total fatty acids.
Body composition | 3 months
  Total body soft tissue composition (fat mass and lean mass) measurements were performed using dual-energy X-ray absorptiometry (DXA) on a stationary fan beam densitometer.
Bone mineral density | 3 months
  The total body bone mineral density (BMD) measurements were performed using dual-energy X-ray absorptiometry (DXA) on a stationary fan beam densitometer.

CONTACTS AND LOCATIONS:
Overall Officials: Ingvild E Graff, PhD, Study Chair — NIFES, postboks 2029 Nordnes, 5815 Bergen, Norway
Locations (1):
- NIFES, Bergen, Norway